CLINICAL TRIAL: NCT00669422
Title: ChemoFx® PRO - A Post-Market Data Collection Study Utilizing Physician Reported Outcomes
Brief Title: ChemoFx® PRO - A Post-Market Data Collection Study
Status: Terminated | Type: Observational
Sponsor: Precision Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: PT-206 ChemoFx® PRO Study
Record Dates: First submitted 2008-04-25; First posted 2008-04-30 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Uterine Neoplasms; Endometrial Cancer; Vaginal Cancer; Vulvar Cancer; Cervical Cancer
Keywords: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer; Uterine Neoplasms; Vulvar Cancer; Endometrial Cancer; Cervical Cancer; Assay; Chemotherapy; Recurrent; Refractory; Persistent; Chemoresponse; Sensitivity; Precision Therapeutics; ChemoFx
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Uterine Neoplasms; Endometrial Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Uterine Cervical Neoplasms; Recurrence; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Leftover tumor cells from the test and pathology slides will be collected and stored to look for potential genetic variations related to drug pathway genes to identify patterns associated with clinical outcome.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will collect patient demographic, oncology history, and physician reported outcome information following the initial round of chemotherapy received after a commercial ChemoFx® Final Report for the generation of hypotheses of potential patient cohorts for further sub-studies.

DETAILED DESCRIPTION:
The traditional treatment course for new cases of many cancers is cytoreductive surgery followed by chemotherapy. Unfortunately, despite high initial response rates to treatment, the majority of patients recur. The use of ineffective chemotherapy can result in unnecessary toxicity and costs, delay of more effective treatment, and the potential for the development of cross-resistance to additional drugs. The ability to individualize therapy by providing the treating physician with ex vivo response information on a panel of drugs should aid in the selection of effective therapy for individual patients, thus resulting in improved outcomes.

ChemoFx® is a drug response marker that quantifies an individual cancer patient's probable tumor response to various chemotherapeutic and biologic agents-providing both sensitivity and resistance information. In a retrospective study, it was demonstrated that patients treated with a regimen that the ChemoFx® test said the patients' cells would be sensitive to, corresponded to a 3 times longer progression free interval.

In the PT-206 ChemoFx PRO® study, patients will be followed through treatment, until the patient progresses or a significant change in chemotherapy occurs. This data will be collected and analyzed to identify potential patient cohorts for the development of hypotheses for future sub-study analysis. Also, tumor pathology slides and excess tumor cells (if available) will be used to characterize common polymorphisms in drug metabolizing enzymes as well as other molecular markers potentially associated with tumor response.

The PT-206 ChemoFx PRO® Study seeks to enroll an estimated 3,000 patients from 150 academic and community-based physicians in the U.S. The patients will be treated with drugs and/or drug combinations based on the medical judgment of the treating physician. This study is not randomized.

ELIGIBILITY:
Inclusion Criteria:

* Patient has been diagnosed with a solid tumor malignancy and their physician has received a final report for ChemoFx® after August 1, 2006
* Chemotherapy must be clinically indicated for treatment of the patient's qualifying disease
* Patient must be at least 18 years of age
* Patient must have signed an IRB approved informed consent form for the data collection study prior to entry of data into the enrollment form in the database.

Exclusion Criteria:

* Patient pathology shows benign pathology for sample submitted
* Patient is not indicated to receive chemotherapy for their disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 3,000 patients from 150 academic and community based physicians in the United States.
  Patients have a confirmed solid tumor malignancy and their tissue specimen has been submitted to Precision Therapeutics, Inc. as part of the patient's medical care
Sampling Method: Non-Probability Sample
Enrollment: 2756 (Actual)
Dates: Start 2006-10; Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To collect physician reported outcomes after the first chemotherapy utilized following the receipt of a final report from ChemoFx® in solid tumor malignancies for the generation of hypotheses for further sub-study. | 24-36 Months depending on Disease Status

SECONDARY OUTCOMES:
Identify possible enhancements of the predictive and prognostic capabilities of the assay through the inclusion of molecular markers. | 24-36 Months depending on Disease Status

CONTACTS AND LOCATIONS:
Locations (67):
- United States (67):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of South Alabama, Mobile, Alabama
  - University of California San Francisco, San Francisco, California
  - Women's Cancer Center of Southern California, Sherman Oaks, California
  - GOA Torrance Memorial, Torrance, California
  - Hartford Hospital, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - South Florida Center for Gynecologic Oncology, Boca Raton, Florida
  - West Coast Gynecologic Oncology, Clearwater, Florida
  - Florida Center for Gynecologic Oncology, Coconut Creek, Florida
  - Comprehensive Gynecologic Oncology, Delray Beach, Florida
  - Caruso and Gates MDs PA, Fort Lauderdale, Florida
  - Florida Gynecologic Oncology, Fort Myers, Florida
  - Gynecologic Oncology Associates, Hollywood, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - South Miami Gynecologic Oncology Group, South Miami, Florida
  - Palm Beach Cancer Institute, West Palm Beach, Florida
  - Southeastern Gynecologic Oncology, LLC, Riverdale, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - The Queens' Medical Center, Honolulu, Hawaii
  - Rush University, Chicago, Illinois
  - NorthShore Medical Group, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - Women's Cancer Center, Covington, Louisiana
  - CHRISTUS Schumpert Health System, Shreveport, Louisiana
  - Sinai Hospital, Baltimore, Maryland
  - Women's Health Specialists, Silver Springs, Maryland
  - UMass Memorial Hospital, Worcester, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Gynecologic Oncology of West Michigan, Grand Rapids, Michigan
  - Mississippi Oncology Associates, Jackson, Mississippi
  - Atlantic Health Systems, Morristown, New Jersey
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Gara M Sommers MD, Teaneck, New Jersey
  - Cooper Health System, Voorhees Township, New Jersey
  - Women's Cancer Care Associates, Albany, New York
  - St. John's Episcopal Hospital, Atlantic Beach, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore LIJ Health System, Manhassett, New York
  - Columbia University Medical Center, New York, New York
  - New York Downtown Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Hope: A Women's Cancer Center, Asheville, North Carolina
  - Blumenthal Cancer Center, Charlotte, North Carolina
  - Presbyterian Gynecologic Oncology, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - North Hanover Regional Medical Center, Wilmington, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - OSU Gynecologic Oncology, Columbus, Ohio
  - Oklahoma Gynecologic Oncology Group, Oklahoma City, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - The Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Women & Infants Hospital of Rhode Island, Providence, Rhode Island
  - Medical University of South Carolina Hospital, Charleston, South Carolina
  - Sandford USD Health System, Sioux Falls, South Dakota
  - Chattanooga Gynecologic Oncology, Chattanooga, Tennessee
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - Thomas W. McDonald MD, Knoxville, Tennessee
  - North Texas Gynecologic Oncology, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - South Texas Gynecologic Oncology, San Antonio, Texas
  - North Virigina Pelvic Surgery Associates, Annandale, Virginia
  - Carilion Clinic Gynecologic Oncology, Roanoke, Virginia
  - Mohammed Ashraf MD, Morgantown, West Virginia
  - Aurora West Allis Medical Center, West Allis, Wisconsin

REFERENCES:
- [Background] Jemal A, Tiwari RC, Murray T, Ghafoor A, Samuels A, Ward E, Feuer EJ, Thun MJ; American Cancer Society. Cancer statistics, 2004. CA Cancer J Clin. 2004 Jan-Feb;54(1):8-29. doi: 10.3322/canjclin.54.1.8. PMID 14974761
- [Background] Ness RB, Wisniewski SR, Eng H, Christopherson W. Cell viability assay for drug testing in ovarian cancer: in vitro kill versus clinical response. Anticancer Res. 2002 Mar-Apr;22(2B):1145-9. PMID 12168915
- [Background] O'Meara AT, Sevin BU. Predictive value of the ATP chemosensitivity assay in epithelial ovarian cancer. Gynecol Oncol. 2001 Nov;83(2):334-42. doi: 10.1006/gyno.2001.6395. PMID 11606094
- [Background] McLeod HL, King CR, Marsh S. Application of pharmacogenomics in the individualization of chemotherapy for gastrointestinal malignancies. Clin Colorectal Cancer. 2004 Jun;4 Suppl 1:S43-7. doi: 10.3816/ccc.2004.s.007. PMID 15212705